CLINICAL TRIAL: NCT04404491
Title: The Third Phase of Immunotherapy and Concurrent Chemoradiotherapy in Patients With Esophageal Cancer Recurrence Was Compared With the Clinical Comparison
Brief Title: Clinical Control Study of Immunotherapy and Concurrent Chemoradiotherapy in Patients With Esophageal Cancer Recurrence
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Henan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITCRTECR
Record Dates: First submitted 2020-05-15; First posted 2020-05-27 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-03

CONDITIONS: Esophageal Malignant Neoplasm, Local Recurrence
Keywords: Carrillizumab; Esophageal cancer recurred; concurrent radiochemotherapy
MeSH Terms: interventions — camrelizumab; Capecitabine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PD-1 and Concurrent chemoradiotherapy (Active Comparator): Camrelizumab: 200mg,d1,15,29,43,57,I.V oxaliplatin：65mg/m2，d1，8，22, 29 capecitabine: 625mg/m2, bid d1-5; q1w, po,6 weeks in total. radiotherapy： 50-50.4Gy ，1.8-2 Gy/d，5d/w.
  Interventions: Drug: Procedural death 1; Drug: Capecitabine; Radiation: Radiotherapy
- placebo and Concurrent chemoradiotherapy (Placebo Comparator): placebo: 200mg,d1,15,29,43,57,I.V oxaliplatin：65mg/m2，d1，8，22, 29 capecitabine: 625mg/m2, bid d1-5; q1w, po,6 weeks in total. radiotherapy： 50-50.4Gy ，1.8-2 Gy/d，5d/w.
  Interventions: Drug: Capecitabine; Radiation: Radiotherapy; Drug: Placebo

INTERVENTIONS:
Drug: Procedural death 1 — 200mg,d1,15,29,43,57,I.V
  Other Names: Camrelizumab
  Arms: PD-1 and Concurrent chemoradiotherapy
Drug: Capecitabine — Capecitabine: 625mg/m2, bid d1-5; q1w, po,6 weeks in total.
  Other Names: Aibin
Radiation: Radiotherapy — radiotherapy： 50-50.4Gy ，1.8-2 Gy/d，5d/w.
  Other Names: Radiation Therapy
Drug: Placebo — placebo: 200mg,d1,15,29,43,57,I.V
  Arms: placebo and Concurrent chemoradiotherapy

SUMMARY:
Esophageal cancer is still a serious threat to human life and health. China in particular. Relapse and metastasis are important causes of treatment failure. Immunotherapy is a new treatment method, which can be used in combination with chemotherapy to improve the therapeutic effect. However, the role of immunotherapy combined with chemoradiotherapy in concurrent chemoradiotherapy of recurrent esophageal cancer has not been clearly studied. Our team will study it in detail.

The purpose of this study was to compare and analyze the effect of Camrelizumab in concurrent chemoradiotherapy of locally recurrent esophageal cancer.

DETAILED DESCRIPTION:
In this study, patients with local recurrence of esophageal carcinoma without distant metastasis were randomly divided into experimental group and control group by Block randomization. In the experimental group, patients with local recurrence were treated with Camrelizumab combined with concurrent chemoradiotherapy. Followed up for 3 years to observe the objective remission rate and disease-free survival. In the control group, patients with local recurrence were treated with placebo combined with concurrent chemoradiotherapy. Followed up for 3 years to observe the objective remission rate and disease-free survival.

ELIGIBILITY:
Inclusion Criteria:

1.Age 18-75 years old, both men and women; 2. Histologically confirmed as esophageal squamous cell carcinoma; 3. Postoperative local recurrence of esophageal cancer (stage II-IVA); 4. According to the evaluation criteria of RECIST 1.1, at least one measurable lesion; 5. ECOG: 0 ～ 1; 6. Expected survival time ≥ 12 weeks; 7. The function of main organs is normal, that is, it meets the following standards: Blood routine examination:a. HB≥90g / L; b.ANC≥1.5 × 109 / L; c.PLT≥80 × 109 / L;3.Biochemical inspection:a.ALB ≥ 30g / L; b. ALT and AST ≤ 2.5ULN; c. TBIL ≤ 1.5ULN; 8. Women of childbearing age should agree to use contraceptive measures (such as intrauterine devices, contraceptives or condoms) during the study period and within 6 months after the end of the study; the serum or urine pregnancy test is negative within 7 days before the study enrollment , and must be a non-lactating patient; males should agree to patients who must use contraception during the study period and within 6 months after the end of the study period; 9. Subjects voluntarily joined the study, signed an informed consent form, had good compliance, and cooperated with follow-up.

Exclusion Criteria:

1. Does not meet the above selection criteria;
2. Patients with distant metastases;
3. Those who are allergic to or metabolic disorders of capecitabine and Camrelizumab;
4. The patient has any active autoimmune disease or has a history of autoimmune disease (such as the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis , Hyperthyroidism; The patient has vitiligo; Asthma has been completely relieved in childhood and can be included without any intervention after adulthood; Patients with asthma requiring medical intervention with bronchodilators cannot be included);
5. The patient is using immunosuppressive agents or systemic hormone therapy to achieve the purpose of immunosuppression (dose> 10mg / day prednisone or other therapeutic hormones), and is still using it within 2 weeks before enrollment; 6. Contraindications to radiotherapy;

7. Severe infections that are active or uncontrolled; 8. Liver diseases such as decompensated liver disease, active hepatitis B (HBV-DNA≥104 copies / ml or 2000IU / ml) or hepatitis C (hepatitis C antibody is positive, and HCV-RNA is higher than the analytical method; 9. Patients whose imaging has shown that the tumor has invaded the important blood vessels or the investigator judges that the tumor is likely to invade the important blood vessels and cause fatal hemorrhage during the follow-up study; 10. Pregnant or lactating women; 11. Patients with other malignant tumors within 5 years (except basal cell carcinoma of the skin and cervical carcinoma in situ); 12. Patients with a history of psychotropic substance abuse who are unable to quit or have mental disorders; 13. Patients who have participated in clinical trials of other drugs within four weeks; 14. According to the judgment of the investigator, there are patients with concomitant diseases that seriously endanger the safety of the patient or affect the completion of the study; 15. The investigator considers it unsuitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Grade 3/4 acute toxicities | 90 days
  rade 3/4 acute toxicities occurred during or within 90 days after CRT
PFS | 1 year
  Progression Free Survival After completion of the CRT

SECONDARY OUTCOMES:
ORR | 16 weeks
  overall remission rate
OS Qol | 1 year
  overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Shegan Gao, M.D,Ph.D, Study Chair — The First Affiliated Hospital of Henan University of Science and Technology

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nakajima T, Ogata T, Nomiya T, Nonaka T, Nakayama Y, Kano K, Maezawa Y, Segami K, Ikeda K, Sato T, Cho H, Yoshikawa T. [Radical Chemoradiotherapy for Recurrent Esophageal Cancer after Curative Esophagectomy]. Gan To Kagaku Ryoho. 2016 Nov;43(12):1564-1566. Japanese. PMID 28133058
- [Background] Zhu LL, Yuan L, Wang H, Ye L, Yao GY, Liu C, Sun NN, Li XJ, Zhai SC, Niu LJ, Zhang JB, Ji HL, Li XM. A Meta-Analysis of Concurrent Chemoradiotherapy for Advanced Esophageal Cancer. PLoS One. 2015 Jun 5;10(6):e0128616. doi: 10.1371/journal.pone.0128616. eCollection 2015. PMID 26046353
- [Background] Jingu K, Umezawa R, Yamamoto T, Matsushita H, Ishikawa Y, Kozumi M, Kubozono M, Takahashi N, Kadoya N, Takeda K. Elective nodal irradiation is not necessary in chemoradiotherapy for postoperative loco-regional recurrent esophageal cancer. Jpn J Clin Oncol. 2017 Mar 1;47(3):200-205. doi: 10.1093/jjco/hyw195. PMID 28031356
- [Background] Fassan M, Cavallin F, Guzzardo V, Kotsafti A, Scarpa M, Cagol M, Chiarion-Sileni V, Maria Saadeh L, Alfieri R, Castagliuolo I, Rugge M, Castoro C, Scarpa M. PD-L1 expression, CD8+ and CD4+ lymphocyte rate are predictive of pathological complete response after neoadjuvant chemoradiotherapy for squamous cell cancer of the thoracic esophagus. Cancer Med. 2019 Oct;8(13):6036-6048. doi: 10.1002/cam4.2359. Epub 2019 Aug 20. PMID 31429521
- [Background] Sato D, Motegi A, Kadota T, Kojima T, Bando H, Shinmura K, Hori K, Yoda Y, Oono Y, Zenda S, Ikematsu H, Akimoto T, Yano T. Therapeutic results of proton beam therapy with concurrent chemotherapy for cT1 esophageal cancer and salvage endoscopic therapy for local recurrence. Esophagus. 2020 Jul;17(3):305-311. doi: 10.1007/s10388-020-00715-y. Epub 2020 Jan 21. PMID 31965362
- [Background] Chen B, Li Q, Li Q, Qiu B, Xi M, Liu M, Hu Y, Zhu Y. Weekly Chemotherapy of 5-Fluorouracil plus Cisplatin Concurrent with Radiotherapy for Esophageal Squamous Cell Carcinoma Patients with Postoperative Locoregional Recurrence: Results from a Phase II Study. Oncologist. 2020 Apr;25(4):308-e625. doi: 10.1634/theoncologist.2019-0931. Epub 2019 Dec 27. PMID 31880371
- [Background] Kelly RJ. Immunotherapy for Esophageal and Gastric Cancer. Am Soc Clin Oncol Educ Book. 2017;37:292-300. doi: 10.1200/EDBK_175231. PMID 28561677
- [Background] Yang H, Wang K, Wang T, Li M, Li B, Li S, Yuan L. The Combination Options and Predictive Biomarkers of PD-1/PD-L1 Inhibitors in Esophageal Cancer. Front Oncol. 2020 Mar 5;10:300. doi: 10.3389/fonc.2020.00300. eCollection 2020. PMID 32195194
- [Background] Kato K, Shah MA, Enzinger P, Bennouna J, Shen L, Adenis A, Sun JM, Cho BC, Ozguroglu M, Kojima T, Kostorov V, Hierro C, Zhu Y, McLean LA, Shah S, Doi T. KEYNOTE-590: Phase III study of first-line chemotherapy with or without pembrolizumab for advanced esophageal cancer. Future Oncol. 2019 Apr;15(10):1057-1066. doi: 10.2217/fon-2018-0609. Epub 2019 Feb 8. PMID 30735435
- [Background] Svensson MC, Borg D, Zhang C, Hedner C, Nodin B, Uhlen M, Mardinoglu A, Leandersson K, Jirstrom K. Expression of PD-L1 and PD-1 in Chemoradiotherapy-Naive Esophageal and Gastric Adenocarcinoma: Relationship With Mismatch Repair Status and Survival. Front Oncol. 2019 Mar 13;9:136. doi: 10.3389/fonc.2019.00136. eCollection 2019. PMID 30931254